CLINICAL TRIAL: NCT02812199
Title: Efficacy of Post-FESS Implantation of Composite Removable Sinus Stent System to Prevent Post-Operative Complications and Revision Surgery
Brief Title: Efficacy of Post-FESS Implantation of Composite Removable Sinus Stent to Prevent Post-Operative Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: STS Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 461001P
Record Dates: First submitted 2016-06-09; First posted 2016-06-24 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- pilot study group 1 (Experimental): Patients in pilot study group 1 will undergo post-FESS bilateral implantation of Composite Removable Sinus Stent into middle meatus. Nasal tampon will be placed to stop bleeding if necessary. Patients in pilot study group scheduled for 6 follow up visits at 1,2,3,4,6 and 12 weeks after implantation and for tampon removal at day 2 - 3 after FESS surgery. Stent will be removed between 14 and 28-day implantation. Before removal adrenaline - lidocaine administration will be used locally to minimize bleeding and cold saline wash applied to induce stent crimping.
  Interventions: Device: Composite Removable Sinus Stent; Drug: adrenaline-lidocaine; Procedure: cold saline wash
- study group 2 (Experimental): Patients in study group 2 will undergo post-FESS bilateral implantation of Composite Removable Sinus Stent into middle meatus. Nasal tampon will be placed to stop bleeding if necessary. Patients in 2nd study group scheduled for 4 follow up visits at 2, 4, 6 and 12 weeks after implantation. Before removal adrenaline - lidocaine administration will be used locally to minimize bleeding and cold saline wash applied to induce stent crimping.
  Interventions: Device: Composite Removable Sinus Stent; Drug: adrenaline-lidocaine; Procedure: cold saline wash
- control group 3 (No Intervention): control group patients will undergo post-FESS bilateral Standard of Care (tampon) placement into middle meatus as standard of care. Frontal tampon will be placed to stop bleeding. Patients in control group scheduled for 3 follow up visits at 2, 6 and 12 weeks after surgery and for tampon removal at day 2 - 3 after FESS surgery.

INTERVENTIONS:
Device: Composite Removable Sinus Stent — Post-FESS bilateral implantation of sinus stent into middle meatus. Nasal tampon will be placed to stop bleeding. Stent will be removed after 14 - 28-day implantation, during self-crimp procedure induced by cold saline flush and safely pulled out. During implantation period patients will be examined endoscopically for inflammation, adhesions and middle turbinate position.
  Arms: pilot study group 1; study group 2
Drug: adrenaline-lidocaine — adrenaline - lidocaine administration to minimize bleeding prior to stent removal (group 1 and group 2)
  Arms: pilot study group 1; study group 2
Procedure: cold saline wash — nasal wash with cold saline prior to stent removal, to induce stent self-crimping.
  Arms: pilot study group 1; study group 2

SUMMARY:
This is a randomized controlled first in man study. Study purpose is to assess safety and efficacy of Composite Removable Stent Composite Stent implantation post-endoscopic sinus surgery in terms of:

* Sinus tissue adhesions
* Middle turbinate lateralization into nasal septum i.e. postoperative opening reduction
* Inflammation

DETAILED DESCRIPTION:
The purpose of this study is to assess Composite Removable Sinus Stent safety and efficacy implantation following FESS surgery compared to standard of care.

At first pilot stage, 3-6 patients will be enrolled to this study. At 2nd stage 19-27 additional patients will be enrolled to this study for statistical assurance.

In study group patients will undergo post-FESS bilateral implantation of Composite Removable Sinus Stent into ethmoid sinus under same anesthesia. Stent is inserted upon low pressure balloon catheter. After reaching target position balloon is inflated and stent deployed and secured. Balloon catheter is deflated and removed. Stent implanted for 14-28-day time period (depending on healing process and therapeutic effect). The stent will be removed upon balloon catheter or using medical grasper, following cooling and self-crimping.

In control group patients will undergo post-FESS bilateral tampon placement into middle meatus as standard of care. Tampon will be removed at day 2-3 post surgery.

Patients in pilot study group (group 1) scheduled for 6 follow up visits at 1,2,3,4,6 and 12 weeks after implantation.

Patients in study group (group 2) scheduled for 4 follow up visits at 2, 4, 6 and 12 weeks after implantation.

Patients in control group (group 3) scheduled for 3 follow up visits at 2, 6 and 12 weeks after surgery. All groups scheduled for tampon removal at day 2 - 3 after ESS surgery (if nessecery) .

During follow up visits patients will be examined for:

* Endoscopic examination of the surgical cavity to assess inflammation, MT position, adhesions and polyposis.

  * Inflammation VAS anchored as o=none and 10cm=severe (significant erythema and edema and/or hypertrophy, and/or polypoid change.
  * Adhesions graded at 5-point scale as none, small but not obstructing, obstructing but easily separated, dense and separation is difficult, severe with complete MT lateralization into lateral nasal wall.
  * MT position graded at 4-point scale as medialized, normal, partially lateralized, and lateralized.
* SNOT - 22 score - taken prior to FESS and at 12 weeks follow up.
* Pain questioner - taken at tampon removal day for group 3 and at stent removal day for groups 1 and 2.

Stent will be removed between 14 and 28-day implantation, during self-crimp procedure induced by cold saline wash and safely pulled out. Stent removal performed after adrenaline-lidocaine administration for minimization of bleeding.

Study Discontinuation

* Patient severe inflammation or pain associated with the stent
* Patient nasal trauma.
* Stent migration
* Nitinol struts exposure as reason for granulation process initiation

ELIGIBILITY:
Inclusion Criteria:

* Male/Female, 18 year or older
* Diagnosis of Recurrent Rhinosinusitis defined as symptomatic inflammation of the sinuse of at least 12 consecutive weeks duration
* CT scan examination with a minimum Lund-MacKay stage of 4 prior to study entry
* Planned Endoscopic Sinus surgery

Exclusion Criteria:

* Pregnant or lactating female
* History of immune deficiency
* Known allergy to Nickel
* Known Polyurethane induced dermatitis
* Cystic Fibrosis
* Severe Polyposis
* Sinonasal tumors
* Ciliary Disfunction
* Acute Sinus Inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Composite Removable Sinus Stent efficacy compared to standard of care | 12 weeks
  The primary objective of this study is to assess Composite Removable Stent efficacy following FESS surgery compared to standard of care, in terms of inflammation, adhesion s, middle turbinate position, and patient symptoms improvement assessed by SNOT-22 questioner.

SECONDARY OUTCOMES:
Pain associated with Composite Stent removal vs. standard of care removal | 4 weeks
  The secondary objective is to assess patients pain associated with Composite Stent removal vs. tampon removal assessed using pain questioner filled in at tampon removal and stent removal days.

OTHER OUTCOMES:
Patient discomfort | 4 weeks
  The objective is to assess patient discomfort resulting from stent implantation vs. standard of care implantation, assessed using discomfort questioner filled at tampon and stent removal days.

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Yaniv, Prof, Principal Investigator — ENT Surgeon
Locations (1):
- Herzliya Medical Center, Herzliya, Israel

IPD SHARING:
Plan to Share IPD: Undecided